CLINICAL TRIAL: NCT04213443
Title: Fetal Growth Pattern in Short Stature Women as a Model for True Intrauterine Growth Restriction Prediction.
Brief Title: Fetal Growth Pattern in Short Stature Women
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Other Study IDs: 0275-19-RMB
Record Dates: First submitted 2019-12-26; First posted 2019-12-30 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Intrauterine Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women of short stature: Women that are under 1.6 meters.
  Interventions: Other: Analysis of a patient registry

INTERVENTIONS:
Other: Analysis of a patient registry — Analysis of a patient registry.

SUMMARY:
Women of short stature tend to be classified regarding fetal growth by the same criteria as women of normal and tall stature. The objective of the following study is to evaluate fetal growth patterns parallel to women's height and try to make conclusions regarding possible definitions of subjective Intra-uterine growth restriction.

DETAILED DESCRIPTION:
Based on a patient registry, women of short stature tend to be classified regarding fetal growth by the same criteria as women of normal and tall stature. The objective of the following study is to evaluate fetal growth patterns parallel to women's height and try to make conclusions regarding possible definitions of subjective Intra-uterine growth restriction.

Informed consent is not required due to the retrospective nature of the study. Patient information including medical, obstetric and general background will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Women under 1.6 meters of height.
* Singleton pregnancy.
* Low risk pregnancy.
* Accurate dating.

Exclusion Criteria:

* Women over 1.6 meters of height.
* Multiple pregnancy.
* High risk pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women
Study Population: Women of short stature under 1.6 meters.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Estimated fetal weight changes. | Up to 1 year from admission.
  Changes in estimated fetal weight during pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam healthcare campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No